CLINICAL TRIAL: NCT04175925
Title: A Double-blind, Placebo-controlled, Randomized, Single and Multiple Ascending Dose Study of the Safety, Pharmacokinetics, and Pharmacodynamics of BMS-986322 in Healthy Participants Including an Open-label Assessment of Food and pH Effects on Relative Bioavailability of BMS-986322
Brief Title: A Study Assessing the Drug Levels, Drug Effects, and Safety of BMS-986322 in Healthy Participants
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Bristol-Myers Squibb (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Sequential | Masking: Quadruple | Purpose: Treatment
Other Study IDs: IM032-007
Record Dates: First submitted 2019-11-13; First posted 2019-11-25 (Actual); Last update posted 2022-05-31 (Actual); Status verified 2022-05

CONDITIONS: Healthy Participants
MeSH Terms: interventions — Famotidine

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (3):
- Part A: BMS-986322 (Experimental)
  Interventions: Drug: BMS-986322; Other: BMS-986322 Placebo
- Part B: BMS-986322 Placebo (Experimental)
  Interventions: Drug: BMS-986322; Other: BMS-986322 Placebo
- Part C: BMS-986322 with famotidine (Experimental)
  Interventions: Drug: BMS-986322; Drug: famotidine

INTERVENTIONS:
Drug: BMS-986322 — Specified Dose on Specified Days
Other: BMS-986322 Placebo — Specified Dose on Specified Days
  Arms: Part A: BMS-986322; Part B: BMS-986322 Placebo
Drug: famotidine — Specified Dose on Specified Days
  Arms: Part C: BMS-986322 with famotidine

SUMMARY:
A Study assessing the drug levels and drug effects of variable doses of BMS-986322 in Healthy Participants compared to a placebo. The study also assesses how BMS-986322 affects the body with food and its acidity levels.

DETAILED DESCRIPTION:
Recruitment temporarily on hold due to COVID-19.

This is a randomized, double-blind, placebo-controlled study which will investigate the safety, tolerability, and PK of single and multiple oral doses of BMS-986322 in healthy subjects. The trial consists of three parts: Part A - a single ascending dose (SAD) safety and pharmacokinetic (PK) evaluation; Part B -a multiple ascending dose (MAD) safety, PK, and pharmacodynamic (PD) evaluation; and Part C - effect of food and pH on PK and safety.

ELIGIBILITY:
Inclusion Criteria:

* Healthy Participant, as determined by no clinically significant deviation from normal in medical history, physical examination, ECGs, and clinical laboratory determinations
* Body mass index (BMI) of 18.0 kg/m^2 to 32.0 kg/m^2, inclusive, and body weight ≥ 50 kg, at screening
* Women and men must agree to follow methods of contraception.

Exclusion Criteria:

* Any significant acute or chronic medical illness
* History of recent infection
* History of allergy to BMS-986322 or other compounds

Other protocol-defined inclusion/exclusion criteria could apply.

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 171 (Actual)
Dates: Start 2019-11-15 (Actual); Primary Completion 2021-07-13 (Actual); Study Completion 2021-07-13 (Actual)

PRIMARY OUTCOMES:
Incidence of Death | up to 12 months
Incidence of Adverse Effects (AEs) | up to 12 months
Incidence of Adverse Events leading to discontinuation | up to 12 months
Incidence of Serious Adverse Events (SAEs) | up to 12 months
Vital signs of body temperature | up to 12 months
Vital signs of blood pressure | up to 12 months
Vital signs of respiratory rate | up to 12 months
Number of Participants with abnormal physical examinations | up to 12 months
Number of clinically significant changes in Electrocardiograms (ECGs) | up to 12 months
Number of clinically significant changes in lab assessment of blood serum | up to 12 months
Number of clinically significant changes in lab assessment of urine | up to 12 months
Number of Clinically significant changes in lab assessment of blood | up to 12 months
Maximum concentration (Cmax) of BMS-986322 in Part C | up to 12 months
Time of maximum concentration (Tmax) of BMS-986322 in Part C | up to 12 months
Terminal elimination rate constant (Lambda_z) of BMS-986322 in Part C | up to 12 months
Terminal elimination half-life (T-Half) of BMS-986322 in Part C | up to 12 months
Area under the plasma concentration-time curve extrapolated to infinity [AUC(INF)] of BMS-986322 in Part C | up to 12 months
Area under the plasma concentration-time curve from time 0 to the last quantifiable concentration [AUC(0-T)] of BMS-986322 in Part C | up to 12 months
Apparent oral clearance (CL/F) of BMS-986322 in Part C | up to 12 months
Apparent volume of distrubution at terminal phase (Vz/F) of BMS-986322 in Part C | up to 12 months

CONTACTS AND LOCATIONS:
Overall Officials: Bristol-Myers Squibb, Study Director — Bristol-Myers Squibb
Locations (1):
- ICON (LPRA) - Lenexa, Lenexa, Kansas, United States

REFERENCES:
- See also: BMS Clinical Trial Information — https://www.bms.com/researchers-and-partners/clinical-trials-and-research.html
- See also: BMS Clinical Trial Patient Recruiting — https://www.bmsstudyconnect.com/s/US/English/USenHome
- See also: Investigator Inquiry Form — https://www.bms.com/researchers-and-partners/clinical-trials-and-research.html
- See also: FDA Safety Alerts and Recalls — https://www.fda.gov/Safety/MedWatch/SafetyInformation/default.htm